CLINICAL TRIAL: NCT04738838
Title: Evaluating Potential Benefits of Intranasal Oxytocin on Undersea Operator Training and Performance: Cold Water Task Performance and Recovery
Brief Title: Oxytocin on Cold Water Task Performance and Recovery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Florida Institute for Human and Machine Cognition (Other)
Collaborators: Office of Naval Research (ONR) (U.S. Federal Agency); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-2020-0002
Record Dates: First submitted 2021-01-06; First posted 2021-02-04 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Cold Exposure
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All will remain blinded until completion of human subjects data collection except the research pharmacist providing intranasal oxytocin or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin Nasal Spray (Experimental): Single dose of intranasal oxytocin (48 IU) prior to testing protocol.
  Interventions: Drug: Oxytocin nasal spray
- Placebo Nasal Spray (Placebo Comparator): Single dose of intranasal treatment with placebo (identical to oxytocin nose spray minus the oxytocin)
  Interventions: Drug: Placebo nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Intranasal treatment with oxytocin via nasal spray (48 IU per dose)
  Other Names: Oxytocin
  Arms: Oxytocin Nasal Spray
Drug: Placebo nasal spray — Intranasal treatment with placebo via nasal spray
  Other Names: Placebo
  Arms: Placebo Nasal Spray

SUMMARY:
Naval Special Warfare (NSW) operators are exposed to a variety of extreme environmental conditions and intense physical demands. In addition to breathing high pressure gases at depth, prolonged cold water immersion and inadequate recovery from sustained physical exertion negatively impact individual and team performance. Biotechnologies that could mitigate the effects of cold as well as support physical recovery represent a significant unmet need for the NSW operational community.

Oxytocin (OT) has a wide range of actions both locally in the brain and peripherally in the body including skeletal muscle. These peripheral effects can be mediated by classic ligand-receptor activation given the abundant expression of the oxytocin receptor in peripheral tissues, along with local expression of OT in peripheral tissues where it is likely to act in an autocrine manner. Exogenous OT via intranasal administration is FDA Investigational New Drug (IND)-approved and has been demonstrated as an easy and safe method to increase circulating OT concentrations that may augment actions on peripheral tissues.

DETAILED DESCRIPTION:
Naval Special Warfare (NSW) operators are exposed to a variety of extreme environmental conditions and intense physical demands. In addition to breathing high pressure gases at depth, prolonged cold water immersion and inadequate recovery from sustained physical exertion negatively impact individual and team performance. Biotechnologies that could mitigate the effects of cold as well as support physical recovery represent a significant unmet need for the NSW operational community.

Oxytocin (OT) has a wide range of actions both locally in the brain and peripherally in the body including skeletal muscle. These peripheral effects can be mediated by classic ligand-receptor activation given the abundant expression of the oxytocin receptor in peripheral tissues, along with local expression of OT in peripheral tissues where it is likely to act in an autocrine manner. Exogenous OT via intranasal administration is FDA Investigational New Drug (IND)-approved and has been demonstrated as an easy and safe method to increase circulating OT concentrations that may augment actions on peripheral tissues.

Cold water operators undergo an extensive and unique set of physical, physiological, and psychological stressors during a mission. In-water transit may exceed 6 hours submerged in cold water, on rebreathers, and in a confined space. During this lengthy transit, operators must maintain vigilance over navigation, vehicle, and life support controls while exposed to the risks of mixed gas or oxygen rebreather diving, alongside hypothermia, dehydration, undernutrition, and other factors that can significantly degrade operator performance. Once the team has reached target, they must be at peak cognitive and physical readiness as they carry out their mission objective. When the mission objective is complete, the operators undertake the lengthy return trip back to their deployed base. Optimized operator cognitive and physical performance is essential throughout all phases of a cold water mission, and safe and tolerable approach to optimizing warfighter performance and resilience will be key for future cold water operations.

Given the potential thermogenic and recovery effects or intranasal OT, we hypothesize that prophylactic OT administration, compared to placebo, will mitigate deficits in mission-relevant performance during and after cold water exposure. For this project we will utilize the ONR Cold Water Performance Task Battery, which was designed based on results from a task analysis combined with input from the cold water operator community. The task battery has been validated for its ability to induce changes in core and peripheral body temperature, manual dexterity, cognitive performance, and physical performance following cold water exposure. Our hypothesis will be tested via one specific aim enrolling N=24 18-39 y/o men by using a rigorous, double-blind, placebo- controlled, within-subjects randomized cross-over trial comparing 48 IU OT vs placebo (saline) in cold water performance and recovery.

Specific Aim 1. To investigate the impact of intranasal OT on cold water task performance and recovery using the ONR Cold Water Performance Task Battery, which includes cold water exposure; cognitive performance testing via oculometric assessment and the Defense Automated Neurobehavioral Assessment (DANA); and physical performance testing via a simulated ruck, ladder climb, and manual dexterity testing.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally skilled swimmers

Exclusion Criteria:

* Smoking/vaping, a history of psychiatric disorders, safety requirements related to the oxytocin administration [hypersensitivity to oxytocin or vasopressin, history of hyponatremia, syndrome of inappropriate antidiuretic hormone secretion, or psychogenic polydipsia, on vasoconstrictors such as desmopressin, pseudoephedrine, or antidiuretic medication, or anti-inflammatory drugs, or muscle relaxants, low sodium and high osmolality levels, excessive smoking, excessive drinking, and significant nasal pathology.

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Cognitive performance assessment score change (code substitution) | Within 3 hours post-treatment
  Changes in code substitution scores as measured by the Defense Automated Neurobehavioral Assessment (DANA). Data will be measured in milliseconds for response time.
Cognitive performance assessment score change (code substitution) | Within 3 hours post-treatment
  Changes in code substitution scores as measured by the Defense Automated Neurobehavioral Assessment (DANA). Data will be measured in number of correct or incorrect responses.
Cognitive performance assessment score change (reaction time) | Within 3 hours post-treatment
  Changes in choice reaction time scores as measured by the Defense Automated Neurobehavioral Assessment (DANA). Data will be measured in milliseconds for response time.
Cognitive performance assessment score change (reaction time) | Within 3 hours post-treatment
  Changes in choice reaction time scores as measured by the Defense Automated Neurobehavioral Assessment (DANA). Data will be measured in number of correct or incorrect responses.
Oculometric assessment score change (saccades) | Within 3 hours post-treatment
  Altered ocular response as measured by the I-Portal Portable Assessment System (i-PAS). Saccades will be monitored and counted throughout the duration of the assessment.
Oculometric assessment score change (blink rate) | Within 3 hours post-treatment
  Altered ocular response as measured by the I-Portal Portable Assessment System (i-PAS). Number of blinks will be counted through the course of the assessment.
Oculometric assessment score change (blink duration) | Within 3 hours post-treatment
  Altered ocular response in blink duration as measured by the I-Portal Portable Assessment System (i-PAS). Blink duration will be measured in milliseconds.

SECONDARY OUTCOMES:
Reduced rating of perceived exertion (RPE) during physical assessment post-cold water exposure | Within 3 hours post-treatment
  Participants will signal on the Borg (6-20) scale for whole body and lower body exertion following their exposure to cold water. Lower on the scale signal a lower level of perceived physical exertion.

OTHER OUTCOMES:
Difference in grip strength in cold water | Within 3 hours post-treatment
  During and after cold water exposure, participants will complete a grip strength assessment through the use of a hand dynamometer. Measurements will be taken in Newtons.
Difference in manual dexterity (underwater knot untying) in cold water | Within 3 hours post-treatment
  During and after cold water exposure, participants will complete a timed underwater knot untying and peg board time trial. Measurement will be recorded in seconds.
Difference in manual dexterity (underwater peg board assessment) in cold water | Within 3 hours post-treatment
  During and after cold water exposure, participants will complete a timed underwater peg board assessment time trial. Measurement will be recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Marcas Bamman, Ph.D., Principal Investigator — Florida Institute for Human and Machine Cognition
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Florida Institute for Human and Machine Cognition, Pensacola, Florida

IPD SHARING:
Plan to Share IPD: No